CLINICAL TRIAL: NCT03803332
Title: A Non-Inferiority Randomized Controlled Clinical Trial Comparing Interpersonal Therapy to Exposure Therapy for PTSD Consequent to Military Sexual Trauma
Brief Title: A Trial Comparing Interpersonal Therapy to Exposure Therapy for PTSD Due to Military Sexual Trauma (MST) in Male and Female Military Personnel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1409015511; W81XWH-16-R-BAA1 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-01-11; First posted 2019-01-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-03

CONDITIONS: PTSD
Keywords: PTSD; Military Sexual Trauma; exposure therapy; interpersonal psychotherapy; treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Military Sexual Trauma | interventions — Implosive Therapy; Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure Therapy (Active Comparator): Participants receive 10 90-minute exposure therapy sessions for PTSD following the treatment procedures as outlined in the standard Prolonged Exposure therapy manual.
  Interventions: Behavioral: Exposure Therapy
- Interpersonal Psychotherapy (Active Comparator): Participants receive 14 weekly 50-minute Interpersonal Psychotherapy sessions focused on the interpersonal sequelae of trauma in current daily life.
  Interventions: Behavioral: Interpersonal Psychotherapy

INTERVENTIONS:
Behavioral: Exposure Therapy — Psychotherapy including imaginal and in vivo exposure for PTSD.
  Other Names: Prolonged Exposure
  Arms: Exposure Therapy
Behavioral: Interpersonal Psychotherapy — Psychotherapy that focuses on the effects of PTSD on current interpersonal functioning.
  Arms: Interpersonal Psychotherapy

SUMMARY:
The purpose of this study is to compare two kinds of therapy for Posttraumatic Stress Disorder (PTSD): exposure therapy (ET) and Interpersonal Psychotherapy (IPT). The results of this study will allow us to see if IPT and ET are equally effective in treating PTSD due to Military Sexual Trauma, with the long-term goal of making PTSD treatment effective for as many people as possible.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Military Sexual Trauma (MST) survivors, with MST defined as actual or threatened sexual violence, from Vietnam era to current Operation Iraqi Freedom/Operation Enduring Freedom/Operation New Dawn
* Diagnosed with PTSD consequent to MST, with a minimum CAPS score > 40
* Medically stable at time of study enrollment (for persons with chronic injuries and that any disability present does not prevent attendance of weekly outpatient therapy sessions)
* Ability to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments
* Stable on psychotropic medication for the prior 60 days

Exclusion Criteria:

* Lifetime or current diagnosis of schizophrenia or other psychotic disorder, bipolar disorder
* Participation in a clinical trial or concurrent evidence-based treatment for MST-related psychiatric conditions or PTSD during the previous 3 months
* Current evidence of significant unstable medical illness or organic brain impairment such that the patient could not attend sessions regularly or complete assessments
* Patients who in the investigator's judgment pose a current homicidal or suicidal risk
* Current or history of substance dependence in the past 90 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Difference in mean Clinician Administered PTSD Scale-5 (CAPS-5) score changes between the Exposure Therapy (ET) and Interpersonal Psychotherapy (IPT) treatment groups from baseline to post-treatment | Baseline, 15 weeks in the IPT condition, 11 weeks in the ET condition
  The CAPS-5 is used for rating the severity of PTSD symptoms. Scores range from 0-80 with higher scores indicating greater PTSD severity
Change in CAPS-5 scores from baseline to post-treatment for the ET treatment group | Baseline, 11 weeks
  The CAPS-5 is used for rating the severity of PTSD symptoms. Scores range from 0-80 with higher scores indicating greater PTSD severity
Change in CAPS-5 scores from baseline to post-treatment for the IPT treatment group | Baseline, 15 weeks
  The CAPS-5 is used for rating the severity of PTSD symptoms. Scores range from 0-80 with higher scores indicating greater PTSD severity

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Difede, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No